CLINICAL TRIAL: NCT04421430
Title: The Effect of Three Different Methods on Venipuncture Pain and Anxiety in Children: Distraction Cards, Virtual Reality, and Buzzy® (Randomized Controlled Trial)
Brief Title: Nonpharmacological Methods for Children in Procedural Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Aynur Aytekin Ozdemir, Associate Professor, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2017-10/9
Record Dates: First submitted 2020-06-03; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Procedural Pain; Procedural Anxiety
Keywords: Anxiety; Children; Nursing; Acute pain management
MeSH Terms: conditions — Pain, Procedural; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants were randomized into the experimental and control groups using a block randomization method. Literature shows that age, gender, and fear are three factors affecting procedural pain and anxiety in children (Ball, Bindler, & Cowen, 2010; Twycross, 2009). Therefore, the variables of age (7-9 and 10-12 years), gender (girls and boys), and fear of procedure (yes and no) were used for block randomization. The blocks were repeated five times in each group (2X2X2X5), and 40 participants were assigned to each. The sealed envelope method was used to randomly assign participants to the groups.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Distraction cards group (Experimental): Distraction cards was applied to the children in this group during the venipuncture procedure.
  Interventions: Other: Distraction cards
- Virtual reality group (Experimental): Virtual reality intervention was applied to the children in this group during the venipuncture procedure.
  Interventions: Other: Virtual reality
- Buzzy® group (Experimental): Buzzy® was applied to the children in this group during the venipuncture procedure.
  Interventions: Other: Buzzy
- Control group (No Intervention): The control group received the routine venipuncture procedure and did not receive any other non-pharmacological intervention.

INTERVENTIONS:
Other: Distraction cards — The distraction cards contain various hidden pictures and patterns which are visible only when looked at carefully. During a procedure, the child is expected to focus on the cards and answer the questions asked about what they see in them. Just before the venipuncture, the researcher showed the distraction cards participants the distraction cards and asked them to check them and then asked them questions about what they saw on the cards and kept asking questions until the end of the venipuncture. The distraction cards intervention and venipuncture were terminated at the same time.
  Other Names: Flippits1, MMJ Labs, Atlanta, Georgia, ABD
  Arms: Distraction cards group
Other: Virtual reality — The virtual reality participants put on the virtual reality glasses and headsets about two minutes before the venipuncture and watched the 3D Dinosaur Animation movie throughout the procedure. The virtual reality intervention and venipuncture were terminated at the same time.
  Arms: Virtual reality group
Other: Buzzy — Buzzy® applies high frequency vibration and concentrated cold at injection site for procedural pain management and distraction before the shot in children and adults. Buzzy® was placed on the injection site (antecubital fossa) of the Buzzy® participants, and cold application and vibration was turned on 60 seconds before the procedure. After the 60 seconds, the nurse moved Buzzy® about 3 cm above the injection site and applied a tourniquet and performed the procedure. Buzzy® was on throughout the procedure. The Buzzy® intervention and venipuncture were terminated at the same time.
  Arms: Buzzy® group

SUMMARY:
The aim of this study was to determine the effect of the distraction cards, virtual reality and Buzzy® methods on venipuncture pain and anxiety in children aged 7-12 years.

DETAILED DESCRIPTION:
The International Guide to Pediatric Anesthesia (Good Practice in Postoperative and Procedural Pain) recommends pharmacological and nonpharmacological methods to effectively manage and prevent acute procedural pain in children. Nonpharmacological methods alone or in combination with pharmacological methods help reduce pain, and therefore, have become popular especially in recent years. For pain management, nonpharmacological methods are easy to use, and cost- and time-effective methods with no side effects. Studies have evaluated a large number of pharmacological and nonpharmacological interventions for procedural pain management in children. However, most of those interventions are not used by healthcare professionals because they are expensive, time-consuming or hard to use. Therefore, easy-to-use, practical, non-invasive, cost-effective, and reusable nonpharmacological methods, such as distraction cards, virtual reality and Buzzy®, can be used especially in acute settings.

ELIGIBILITY:
Inclusion Criteria:

* Due to undergo venipuncture for blood testing
* Suitable for venipuncture at antecubital location using a 21 Gauge X 1.5 inch needle
* Due to undergo venipuncture under the same environmental conditions (phlebotomy seat, heat, light, noise, etc.)
* Due to undergo venipuncture at the first attempt

Exclusion Criteria:

Children;

* had chronic diseases
* had neuro-developmentally delayed
* had visual, audio, or speech impairments
* were hospital stay for treatment
* had a history of sedative, analgesic or narcotic use within 24 hours before admission

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-08-14 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Through painful procedure completion, an average of 10 minutes
  The VAS is used to measure and monitor pain intensity. VAS is a 10 cm or 100 mm long horizontal or vertical line with anchor statements "no pain or pain at its least" at the left-most end and "unbearable pain or worst pain imaginable" at the right-most end. The participant is asked to mark a point on the line that best represents their pain level. The VAS score is determined by measuring (in cm) the distance of the mark from the left end of the line. VAS is an easy-to-understand and easy-to-measure scale for children aged 7 and over.
Wong-Baker FACES Pain Rating Scale (WB-FACES) | Through painful procedure completion, an average of 10 minutes
  The WB-FACES was developed by Wong and Baker in 1981 and revised in 1983. The scale is used to diagnose pain in children aged 3-18 years. It consists of six facial expressions, each one representing an increasing degree of pain scored on a scale 0 to 5 from left to right (0 = very happy/no pain, 5 = the worst pain imaginable). The first face is a happy face representing "no pain" (0) while the last face is a crying face representing "the worst pain imaginable" (5). Higher scores indicate low pain tolerance. Participants are asked to choose the facial expression that best represents their pain.
Children's Fear Scale (CFS) | Through painful procedure completion, an average of 10 minutes
  The CFS was developed by McMurtry et al. (2011) to measure fear and anxiety in children. It consists of five facial expressions that represent a range from neutral (0) to extreme fear (4). Both researchers and family members can use the CFS to measure fear and anxiety in children before and during procedures

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Aytekin Ozdemir, PhD, Principal Investigator — Istanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared after the article is published.

REFERENCES:
- [Background] Ball, J. W., Bindler, R. C., &Cowen, K. J. (2010). Child Health Nursing: Partnering withak Children and Families. (2 th ed.) London: Pearson Education (Chapter 2).
- [Background] Twycross A. (2009). Managing pain in children. In: Dowden, S. J., & Bruce, E., (eds.). A Clinical Guide (pp. 42-49). New Jersey: Blackwell Publishing Ltd.
- [Background] Wong DL, Baker CM. Pain in children: comparison of assessment scales. Pediatr Nurs. 1988 Jan-Feb;14(1):9-17. No abstract available. PMID 3344163
- [Background] McMurtry CM, Noel M, Chambers CT, McGrath PJ. Children's fear during procedural pain: preliminary investigation of the Children's Fear Scale. Health Psychol. 2011 Nov;30(6):780-8. doi: 10.1037/a0024817. Epub 2011 Aug 1. PMID 21806301
- [Derived] Erdogan B, Aytekin Ozdemir A. The Effect of Three Different Methods on Venipuncture Pain and Anxiety in Children: Distraction Cards, Virtual Reality, and Buzzy(R) (Randomized Controlled Trial). J Pediatr Nurs. 2021 May-Jun;58:e54-e62. doi: 10.1016/j.pedn.2021.01.001. Epub 2021 Jan 21. PMID 33485746